CLINICAL TRIAL: NCT03223298
Title: Comparison of Botulinum Toxin Versus Placebo Injections to Temporalis and Masseter Muscles in the Management of Myofascial Pain Disorder: A Randomized Clinical Trial
Brief Title: Botulinum Toxin Versus Placebo Injections to Temporalis and Masseter Muscles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other); Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1607017383
Record Dates: First submitted 2017-07-11; First posted 2017-07-21 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Pain, Head; Pain Syndrome; Temporomandibular Disorder; Myofascial Pain Syndrome; Myofascial Pain
Keywords: Myofascial Pain; Myofascial Pain Disorder; Maxillofacial Pain; Masseter Muscle; Temporalis Muscle; Botulinum Toxin
MeSH Terms: conditions — Headache; Somatoform Disorders; Temporomandibular Joint Disorders; Myofascial Pain Syndromes | interventions — Botulinum Toxins, Type A; Idoxuridine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly allocated to one of two treatment arms (injection of botulinum versus placebo). Blocked randomization will be performed at each of the participating sites. They will be stratified based on study site.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be carried out by the biostatistics team at Weill Cornell. This will provide assurance that there will be equal patient allocation to both study arms, at each participating site, in the event that the target sample size is not reached. The list will be maintained by the investigational pharmacy. A designated research assistant will be identified at each site to prepare the interventional medication (botulinum versus normal saline). The identity of the agent injected will be unknown to the surgeon as the agent will be drawn up by an assistant in a masked syringe immediately prior to each procedure and labeled with the patient's identifier. Only one assistant at each site will know the identity of the agents during the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum Toxin Type A (Experimental): The intramuscular injections will be performed with the patient awake in the oral and maxillofacial surgery clinic. Three injection sites into bilateral masseter muscles and two injection sites into bilateral temporalis muscles will be identified by having the patient clench. The sites will be marked with a surgical pen prior to injections. The skin at the injection sites will be cleaned with an alcohol swab. Via a 1cc TB syringe and a 30-gauge needle, the subject will then receive 100 units of reconstituted botulinum toxin A. 37.5 units will be injected into each masseter muscle and 12.5 units into each temporalis muscle. A written post-operative instruction sheet will be provided to all patients.
  Interventions: Drug: Botulinum toxin type A
- 0.9% Sodium Chloride Injection (Placebo Comparator): The intramuscular injections will be performed with the patient awake in the oral and maxillofacial surgery clinic. Three injection sites into bilateral masseter muscles and two injection sites into bilateral temporalis muscles will be identified by having the patient clench. The sites will be marked with a surgical pen prior to injections. The skin at the injection sites will be cleaned with an alcohol swab. Via a 1cc TB syringe and a 30-gauge needle, the subject will then receive unpreserved 0.9% sodium chloride. A written post-operative instruction sheet will be provided to all patients.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Botulinum toxin type A — 37.5 units injected into each masseter muscle and 12.5 units into each temporalis muscle
  Other Names: Botulinum; Botox; Allergan; Botulinum Toxin A
  Arms: Botulinum Toxin Type A
Drug: 0.9% Sodium Chloride Injection — 1cc syringe
  Other Names: Saline; Placebo
  Arms: 0.9% Sodium Chloride Injection

SUMMARY:
This study aims to determine whether the injection of botulinum toxin A or placebo (unpreserved 0.9% sodium chloride) into the masseter and temporalis muscles provides pain relief and improved jaw function in those who suffer from myofascial pain disorder. The study hypothesis is that botulinum toxin A injection is superior to placebo. The specific research questions are:

1. Is the injection of botulinum toxin A superior to placebo for the improvement in pain?
2. Is the injection of botulinum toxin A superior to placebo for the improvement in function or quality of life (QOL)?
3. Are there any adverse effects that result from injection of botulinum toxin A or placebo into the masseters and temporalis muscles? Limited data exists to support the use of botulinum toxin A in the management of myofascial pain disorder of the masticatory region. Botulinum toxin A is not FDA approved for intra-muscular injection within the masticatory region. Its use in the masticatory region is considered off-label but performed without significant known complications. This study will provide the opportunity to quantitate and qualitate any complications in a large prospective sample of patients.

DETAILED DESCRIPTION:
Myofascial pain is classically used to describe pain experienced in the masticatory muscles and its associated structures (Freund 1999). It afflicts nearly 10% of Americans (Freund 2000). There have been many described treatments such as the use of oral appliances, non-steroidal anti-inflammatory medications, physiotherapy, behavioral therapy and counseling, acupuncture, and botulinum toxin injections (Freund 2000). However, no single treatment has been found to be significantly superior to the others (Freund 2000).

This is a randomized, double-blind, placebo-controlled multicenter study. Subjects will be recruited from the divisions of Oral and Maxillofacial Surgery from all sites. Patients aged 18-65 years with myofascial pain involving the temporalis and masseters are eligible to enter the study. A complete history and physical examination will be performed for all patients in order to make an accurate diagnosis. The research diagnostic criteria (RDC/TMD) will be used to assign a diagnosis of myofascial pain of the masticatory region. All investigators and site-specific data collectors will be trained and calibrated in physical examination techniques and data collection to ensure uniformity between sites. Patients will complete a visual analog scale regarding pain during their screening appointment. To participate in the study, the subject must have greater than or equal to 3.5/10 on the visual analog scale of pain. Informed written consent will be obtained from all patients. Any patient lacking the capacity to make medical decisions will be excluded from the study, although they will be treated as deemed medically necessary. Consent will be written at the sixth grade level, and all potential subjects will be asked to verbally repeat the purpose, methods, and required follow-up to ensure adequate understanding.

The site specific PI will educate fellow faculty and referring departments that the study is enrolling new subjects, advertising is anticipated, and referring physicians will not receive any financial compensation. The intent is to enroll a total of 110 subjects from all sites. The study participants will be reimbursed $25 per treatment visit for their participation.

Previous studies have demonstrated a reduction of pain as indicated on the visual analogue scale of 45% and 32% with the use of intramuscular botulinum toxin A injections into masseter and temporalis (Freund 1999, Guarda-Nardini 2012). Von Lindern et. al. found a mean reduction of 3.2 points on a visual analog scale in the verum group. Based on the preliminary data and the sample size calculations estimating a difference in mean pre-post VAS change between groups of 1 point or greater (on a scale of 1-10), we plan to enroll a total of 110 subjects. With 50 patients in the botulinum toxin A injection group and 50 patients in the placebo group (N=100), the study will have more than 90% power to detect a difference in mean in pre-post change between groups of 1.0 point or greater on VAS, using a two-sided t-test and assuming a standard deviation of 1.5 for the mean difference. This calculation allows for 10% attrition rate. An intent-to-treat design will be followed and all subjects will have scheduled outcome evaluations until the end of the study, death of the subject, or subject refusal. Subjects will be withdrawn from their randomly assigned treatment for considerations of subject safety only.

Descriptive statistics including mean, standard deviation, median, range, frequency, and percent will be calculated for the entire cohort as well as by the study arm (botulinum toxin A and unpreserved 0.9% sodium chloride) to assess the results of randomization and identify potential confounders. The primary analyses of the data will be performed according to subjects' original treatment assignment (i.e., intention-to-treat analyses) and the inclusion of all data from all subjects randomized in the final analysis. To assess the primary endpoint of improvement of pain on a visual analog scale (VAS) between pre-op, 1, 2, and month post-op, and 3 months post-op, a repeated measure of analysis of variance will be performed with one between subject factor (botulinum toxin A versus placebo) and one within subject factor (time). This analysis will also be used for the secondary endpoints: function (MIO/jaw limitation scale) and quality of life (SF12). In the event of significant loss to follow-up, we will explore the use of a linear mixed model to assess the independent effect of the study group on VAS over the study visits. The paired t-test, or the signed-rank test as appropriate, will be used to assess change in pain, function, and QOL between pairs of relevant time points for both study arms. To assess the difference in proportion of adverse events between the botulinum toxin A and placebo groups, either the chi-square or Fisher's exact test will be used, as appropriate. All p-values will be two-sided with statistical significance evaluated at the 0.05 alpha level. Ninety-five percent confidence intervals (95% CI) will be calculated to assess the precision of the obtained estimates. All analyses will be performed in SAS Version 9.4 (SAS Institute Inc., Cary, NC). Note: This section was drafted in conjunction with Dr. Paul Christos and Gulce Askin, MPH in the Division of Biostatistics and Epidemiology, Department of Healthcare Policy and Research. They will be aiding in protocol design and development, data management, study implementation, study monitoring, and data analysis and reporting.

Adverse events will be reported to the Data and Safety Monitoring Board every six months. The participants will be provided with the phone number of the primary investigator and co-investigators for use in reporting any adverse events. The study participants will also be questioned at one, two, and and three months post-treatment for the occurrence of any adverse events. The report of any such events will provide details including severity, relationship to treatment, onset, duration, and outcome. The Data and Safety Monitoring Board will regularly review these reports, and should any trend develop that suggests significant adverse outcomes, the study will be discontinued. If any serious adverse events occur (death, life-threatening, those involving prolonged hospitalization or disability), the independent study monitor, other study sites, IRBs, and DSMB will be notified with 24 hours in the case of death or 72 hours in the event of other serious adverse events.

IRB approval for this study is currently in process (assigned protocol number 1607017383). Pending approval from the IRB for each involved site, research investigators will honor their responsibility to safeguard the rights and welfare of individuals who are or may become subjects of research. Investigators will also maintain compliance with Department of Health and Human Services regulations. All requirements and determinations made by the IRB will be followed to minimize unnecessary risks to subjects. The investigators will abide by procedures consistent with sound research design. Botulinum toxin A is currently not FDA approved for use in myofascial pain disorder of the masticatory region. If the IRB deems its use a "subject risk," an application for investigational new drug (IND) will be submitted to the FDA under the research or noncommercial category. This requirement is not anticipated given the routine use of botulinum toxin A, previous studies demonstrating benefit with minimal risk, and its existing FDA approval for use in the masseter and temporalis muscles for orofacial dystonia/dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Ability to give informed consent
* Myofascial pain of masticatory muscles as defined according to the RDC/TMD criteria
* Baseline pain measured by the subject ≥3.5/10 on visual analog scale

Exclusion Criteria:

* Baseline pain measured by the subject <3.5/10 on visual analog scale
* Central/Neuropathic pain disorder affecting the masticatory muscles
* Temporomandibular Joint Arthralgia that is more severe than the myofascial pain disorder affecting the masticatory muscles
* Previous Temporomandibular Joint Surgery
* Systemic arthropathies
* Fibromyalgia
* Allergy to study medications
* Traumatic injury of masticatory muscles or temporomandibular joint within last 12 months
* Mandibular fracture within last 12 months
* Pregnancy or breast feeding
* Cervical radiculopathy or surgery
* Prior botox injection in the masticatory muscles
* Initiation of additional treatment of MPD within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn S Reeve, DMD, Principal Investigator — Weill Medical College of Cornell University; Michael Miloro, DMD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Weill Cornell Medical College - NewYork-Presbyterian Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botulinum Toxin A for Myofascial Pain Syndrome: A Review of the Clinical Effectiveness [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2014 Sep 22. Available from http://www.ncbi.nlm.nih.gov/books/NBK253364/ PMID 25392894
- [Background] Freund B, Schwartz M, Symington JM. Botulinum toxin: new treatment for temporomandibular disorders. Br J Oral Maxillofac Surg. 2000 Oct;38(5):466-71. doi: 10.1054/bjom.1999.0238. PMID 11010775
- [Background] Freund B, Schwartz M, Symington JM. The use of botulinum toxin for the treatment of temporomandibular disorders: preliminary findings. J Oral Maxillofac Surg. 1999 Aug;57(8):916-20; discussion 920-1. doi: 10.1016/s0278-2391(99)90007-1. PMID 10437718
- [Background] Guarda-Nardini L, Stecco A, Stecco C, Masiero S, Manfredini D. Myofascial pain of the jaw muscles: comparison of short-term effectiveness of botulinum toxin injections and fascial manipulation technique. Cranio. 2012 Apr;30(2):95-102. doi: 10.1179/crn.2012.014. PMID 22606852
- [Background] Soares A, Andriolo RB, Atallah AN, da Silva EM. Botulinum toxin for myofascial pain syndromes in adults. Cochrane Database Syst Rev. 2014 Jul 25;2014(7):CD007533. doi: 10.1002/14651858.CD007533.pub3. PMID 25062018
- [Background] von Lindern JJ, Niederhagen B, Berge S, Appel T. Type A botulinum toxin in the treatment of chronic facial pain associated with masticatory hyperactivity. J Oral Maxillofac Surg. 2003 Jul;61(7):774-8. doi: 10.1016/s0278-2391(03)00153-8. PMID 12856249
- [Derived] Reeve GS, Insel O, Thomas C, Houle AN, Miloro M. Does the Use of Botulinum Toxin in Treatment of Myofascial Pain Disorder of the Masseters and Temporalis Muscles Reduce Pain, Improve Function, or Enhance Quality of Life? J Oral Maxillofac Surg. 2024 Apr;82(4):393-401. doi: 10.1016/j.joms.2023.12.014. Epub 2023 Dec 28. PMID 38228287

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride Injection
Started | 38 | 37
Pre-op | 38 | 37
Month 1 Post-op | 34 | 32
Month 2 Post-op | 22 | 28
Month 3 Post-op | 23 | 27
Completed | 23 | 27
Not Completed | 15 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride Injection | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 37 | 75
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 61
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian / Pacific Islander | 9 | 4 | 13
  Black or African American | 0 | 2 | 2
  Hispanic or Latino | 6 | 7 | 13
  White | 22 | 22 | 44
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Jaw Pain as Reported by Patient on Visual Analog Scale (VAS)
Description: Visual Analog Scale ranging from "no pain (0)" to "pain as bad as it could possibly be (100)"
Time Frame: Pre-intervention, Change at 1 month post-intervention, Change at 2 months post-intervention, Change at 3 months post-intervention
Population: Patient retention varied per time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride Injection
Number analyzed (Participants) | 38 | 37
score on a scale
  Pre-intervention | 58 (15) | 54 (14)
  Change at 1 months post-intervention: number analyzed (Participants) | 34 | 32
  Change at 1 months post-intervention | -19 (24) | -14 (23)
  Change at 2 months post-intervention: number analyzed (Participants) | 22 | 28
  Change at 2 months post-intervention | -18 (24) | -18 (23)
  Change at 3 months post-intervention: number analyzed (Participants) | 23 | 27
  Change at 3 months post-intervention | -17 (22) | -16 (23)
Statistical Analysis 1: Comparison: Botulinum Toxin Type A vs 0.9% Sodium Chloride Injection; 3-month mean change (from pre-op) in Jaw Pain compared between the Botox group and Placebo group; Test type: Superiority; p = 0.80, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Jaw Function as Measured by Jaw Function Limitation Scale
Description: A series of yes or no questions to determine what activities a patient's jaw problem prevents or limits them from doing. A high score of 7 indicates severe jaw limitation, a low score of 0 indicates no jaw limitation.
Time Frame: Pre-intervention, 1 month post-intervention, 2 months post-intervention, 3 months post-intervention
Population: Patient retention varied per time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride Injection
Number analyzed (Participants) | 38 | 37
score on a scale
  Pre-intervention | 0.38 [0.25 to 0.63] | 0.38 [0.25 to 0.50]
  1 month post-intervention: number analyzed (Participants) | 34 | 32
  1 month post-intervention | 0.38 [0.13 to 0.38] | 0.25 [0.13 to 0.38]
  2 months post-intervention: number analyzed (Participants) | 22 | 28
  2 months post-intervention | 0.25 [0.25 to 0.50] | 0.25 [0.13 to 0.38]
  3 months post-intervention: number analyzed (Participants) | 23 | 27
  3 months post-intervention | 0.25 [0.13 to 0.44] | 0.25 [0.06 to 0.38]
Statistical Analysis 1: Comparison: Botulinum Toxin Type A vs 0.9% Sodium Chloride Injection; 3-month mean Jaw Function Limitation Scale score compared between Botox group and placebo group; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Jaw Function as Measured by Maximum Interincisal Opening (MIO)
Description: Mouth opening measurements in mm both when patient is in pain and not in pain. This measurement is taken from the maxillary central incisor to mandibular central incisor.
Time Frame: as for outcome 1
Population: Patient retention varied per time point
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride Injection
Number analyzed (Participants) | 38 | 37
mm
  MIO with Pain: Pre-intervention | 41 (7) | 42 (8)
  MIO without Pain: Pre-Intervention | 34 (7) | 34 (10)
  Change in MIO with Pain at 1-month post-intervention: number analyzed (Participants) | 34 | 32
  Change in MIO with Pain at 1-month post-intervention | 0 (5) | 2 (6)
  Change in MIO without Pain at 1-month post-intervention: number analyzed (Participants) | 34 | 32
  Change in MIO without Pain at 1-month post-intervention | 1 (6) | 4 (8)
  Change in MIO with Pain at 2-months post-intervention: number analyzed (Participants) | 22 | 28
  Change in MIO with Pain at 2-months post-intervention | -1 (7) | 1 (7)
  Change in MIO without Pain at 2-months post-intervention: number analyzed (Participants) | 22 | 28
  Change in MIO without Pain at 2-months post-intervention | -1 (8) | 3 (8)
  Change in MIO with Pain at 3-months post-intervention: number analyzed (Participants) | 23 | 27
  Change in MIO with Pain at 3-months post-intervention | -1 (5) | 1 (8)
  Change in MIO without Pain at 3-months post-intervention: number analyzed (Participants) | 23 | 27
  Change in MIO without Pain at 3-months post-intervention | 2 (8) | 4 (8)
Statistical Analysis 1: Comparison: Botulinum Toxin Type A vs 0.9% Sodium Chloride Injection; Change in MIO with Pain at 3-months post-intervention compared between Botox group and Placebo group; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Botulinum Toxin Type A vs 0.9% Sodium Chloride Injection; Change in MIO without Pain at 3-months post-intervention compared between Botox group and Placebo group; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Objectively Assessed Quality of Life as Measured by Short Form 36
Description: Short Form 36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are utilized for routine monitoring and assessment of care outcomes in adult patients. A high score of 100 on this survey indicates the patient is self-reporting a high quality-of-life, a low score of 0 indicates a low quality-of-life.
Time Frame: as for outcome 1
Population: Patient retention varied per time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride Injection
Number analyzed (Participants) | 38 | 37
score on a scale
  Pre-intervention - Physical Functioning Score | 100 [95 to 100] | 100 [90 to 100]
  Change at 1 month post intervention - Physical Functioning Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - Physical Functioning Score | 0 [0 to 0] | 0 [0 to 0]
  Change at 2 months post-intervention - Physical Functioning Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post-intervention - Physical Functioning Score | 0 [0 to 0] | 0 [0 to 5]
  Change at 3 months post-intervention - Physical Functioning Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post-intervention - Physical Functioning Score | 0 [0 to 0] | 0 [0 to 2]
  Pre-intervention - Role Limitations - Physical Health Score | 100 [75 to 100] | 100 [50 to 100]
  Change at 1 month post intervention - Role Limitations - Physical Health Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - Role Limitations - Physical Health Score | 0 [0 to 0] | 0 [0 to 0]
  Change at 2 months post intervention - Role Limitations- Physical Health Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post intervention - Role Limitations- Physical Health Score | 0 [0 to 0] | 0 [0 to 0]
  Change at 3 months post intervention - Role Limitations - Physical Health Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post intervention - Role Limitations - Physical Health Score | 0 [0 to 0] | 0 [0 to 25]
  Pre-intervention - Role Limitations - Emotional Score | 100 [67 to 100] | 100 [33 to 100]
  Change at 1 month post intervention - Role Limitations - Emotional Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - Role Limitations - Emotional Score | 0 [0 to 0] | 0 [0 to 33]
  Change at 2 months post intervention - Role Limitations - Emotional Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post intervention - Role Limitations - Emotional Score | 0 [0 to 0] | 0 [0 to 33]
  Change at 3 months post intervention - Role Limitations - Emotional Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post intervention - Role Limitations - Emotional Score | 0 [0 to 0] | 0 [-33 to 33]
  Pre-intervention - Energy/Fatigue Score | 50 [45 to 70] | 60 [35 to 65]
  Change at 1 month post intervention - Energy/Fatigue Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - Energy/Fatigue Score | 5 [-4 to 10] | 0 [-5 to 11]
  Change at 2 months post intervention - Energy/Fatigue Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post intervention - Energy/Fatigue Score | 2 [-4 to 15] | 5 [-5 to 11]
  Change at 3 months post intervention - Energy/Fatigue Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post intervention - Energy/Fatigue Score | 5 [-2 to 10] | 0 [-5 to 15]
  Pre-intervention - Emotional Well-Being Score | 76 [64 to 84] | 68 [52 to 84]
  Change at 1 month post intervention - Emotional Well-Being Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - Emotional Well-Being Score | 2 [0 to 8] | 4 [-4 to 13]
  Change at 2 months post intervention - Emotional Well-Being Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post intervention - Emotional Well-Being Score | 4 [0 to 8] | 8 [-1 to 13]
  Change at 3 months post intervention - Emotional Well-Being Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post intervention - Emotional Well-Being Score | 4 [-6 to 6] | 4 [0 to 14]
  Pre-intervention - Social Functioning Score | 100 [75 to 100] | 88 [50 to 100]
  Change at 1 month post intervention - Social Functioning Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - Social Functioning Score | 0 [-12 to 12] | 0 [-3 to 12]
  Change at 2 months post intervention - Social Functioning Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post intervention - Social Functioning Score | 0 [0 to 12] | 0 [0 to 16]
  Change at 3 months post intervention - Social Functioning Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post intervention - Social Functioning Score | 0 [-25 to 12] | 0 [-12 to 12]
  Pre-intervention - Pain Score | 78 [58 to 90] | 58 [55 to 78]
  Change at 1 month post intervention - Pain Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - Pain Score | 0 [-2 to 12] | 10 [0 to 25]
  Change at 2 months post intervention - Pain Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post intervention - Pain Score | 0 [-10 to 18] | 11 [0 to 22]
  Change at 3 months post intervention - Pain Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post intervention - Pain Score | 0 [-5 to 18] | 10 [-6 to 32]
  Pre-intervention - General Health Score | 75 [60 to 85] | 70 [55 to 85]
  Change at 1 month post intervention - General Health Score: number analyzed (Participants) | 34 | 32
  Change at 1 month post intervention - General Health Score | 0 [-5 to 10] | 0 [-1 to 10]
  Change at 2 months post intervention - General Health Score: number analyzed (Participants) | 22 | 28
  Change at 2 months post intervention - General Health Score | 2 [0 to 10] | 5 [-5 to 6]
  Change at 3 months post intervention - General Health Score: number analyzed (Participants) | 23 | 27
  Change at 3 months post intervention - General Health Score | 0 [-5 to 5] | 5 [-5 to 10]
Statistical Analysis 1: Comparison: Botulinum Toxin Type A vs 0.9% Sodium Chloride Injection; Mean change at 3 months post intervention - General Health Score, compared between Botox group and Placebo group; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Botulinum Toxin Type A | 0.9% Sodium Chloride Injection
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 6/38 | 3/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin Type A (N=38) | 0.9% Sodium Chloride Injection (N=37)
Increase in pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) — Mild pain and/or increase in pain
Headaches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Increased frequency of headaches
Mild weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild right side buccal branch weakness that is improving-not bothersome to patient, able to animate bilaterally
Masseter tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — None, having some masseter tenderness over last week
Ecchymosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Ecchymosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03223298/Prot_SAP_000.pdf